CLINICAL TRIAL: NCT06430619
Title: New Criteria for Classifying Acute Respiratory Distress Syndrome Severity Using a Machine Learning Approach: Novel Oxygenation and Saturation Indices
Brief Title: Can Novel Oxygenation Indices Guide the Diagnosis of Acute Respiratory Distress Syndrome
Status: Completed | Type: Observational
Sponsor: Başakşehir Çam & Sakura City Hospital (Other Government)
Collaborators: SBÜ Dr. Sadi Konuk Eğitim ve Araştırma Hastanesi (Other)
Responsible Party: Principal Investigator, Furkan Tontu, Doctor of Anesthesiology and Reanimation, Başakşehir Çam & Sakura City Hospital
Other Study IDs: 2024-40
Record Dates: First submitted 2024-05-09; First posted 2024-05-28 (Actual); Last update posted 2024-05-28 (Actual); Status verified 2024-05

CONDITIONS: Respiratory Distress Syndrome, Adult
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients diagnosed with Acute Respiratory Distress Syndrome (ARDS) according to Berlin criteria: The oxygenation indexes of the patients will be measured and the effectiveness of these indexes in diagnosing ARDS will be compared.

SUMMARY:
This study aims to determine the cut-off values of the new oxygenation indices and further investigate their capabilities in diagnosing ARDS and predicting its severity in ICU. Additionally, the investigators aim to compare these results with conventional oxygenation and saturation indices.

DETAILED DESCRIPTION:
Recent studies have shown that mechanical power (MP) values below 17 J/min and driving pressure (DP) values below 15 cmH2O reduce intensive care unit (ICU) mortality. Asar et al. have introduced six new oxygenation indices utilizing MP and DP instead of Pmean (OSI-MPtot, OI-MPtot, OSI-ΔPinsp, OI-ΔPinsp, OSI-MPdyn, OI-MPdyn). They compared the predictive abilities of these new indices for ICU mortality in Covid-ARDS (C-ARDS) patients with conventional oxygenation indices (P/F, SpO2/FiO2, OI, OSI, PaO2/(FiO2xPEEP), and SpO2/FiO2xPEEP). OI-ΔPinsp, OSI-ΔPinsp, and OSI-MPdyn indices exhibited the highest predictive power for ICU mortality. However, cut-off values for the diagnosis and severity determination (mild, moderate, and severe) of ARDS patients have not been investigated.

In this study, our objective is to determine the cut-off values of the new oxygenation indices and further investigate their capabilities in diagnosing ARDS and predicting its severity in ICU. Additionally, the investigators aim to compare these results with conventional oxygenation and saturation indices.

ELIGIBILITY:
Inclusion Criteria:

1. Patients admitted to intensive care units diagnosed with ARDS / C-ARDS according to the Berlin criteria.
2. Adult patients aged between 18 and 80 years

Exclusion Criteria:

1. Patients under the age of 18
2. Pregnant patients
3. Patients without ARDS
4. Patients with missing data
5. Patients transferred to another hospital
6. Patients discharged from the ICU within 72 hours
7. Patients receiving extracorporeal membrane oxygenation (ECMO) support.
8. Patients were on mechanical ventilation for less than 24 hours

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to the intensive care unit of Istanbul Bakırköy Dr. Sadi Konuk Training and Research Hospital with a preliminary diagnosis of ARDS/C-ARDS between June 01, 2012, and February 01, 2024
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Actual)
Dates: Start 2012-06-01 (Actual); Primary Completion 2024-02-01 (Actual); Study Completion 2024-05-01 (Actual)

PRIMARY OUTCOMES:
Oxygenation indices | During 28 days in the intensive care unit
  It was aimed to compare the oxygenation indexes of the patients. It will be examined which of these indices is more effective in diagnosing ARDS.

SECONDARY OUTCOMES:
Other parameters | During 28 days in the intensive care unit
  It was aimed to compare the sequential organ failure assessment scores of the patients.
  Score ranges from 0 (best outcome) to 24 (worst outcome) points.
acute physiology and chronic health evaluation-II | During 28 days in the intensive care unit
  It was aimed to compare the acute physiology and chronic health evaluation-II scores of the patients.
  Score ranges from 0 (best outcome) to 71 (worst outcome) points.
Charlson comorbidity index scores | During 28 days in the intensive care unit
  It was aimed to compare the Charlson comorbidity index scores of the patients. Based on the Charlson comorbidity index score, the severity of comorbidity was categorized into three grades: mild, with Charlson comorbidity index scores of 1-2; moderate, with Charlson comorbidity index scores of 3-4; and severe, with Charlson comorbidity index scores ≥5.
Other parameters | During 28 days in the intensive care unit
  It was aimed to compare the Charlson comorbidity index of the patients.
arterial blood gas parameters | During 28 days in the intensive care unit
  It was aimed to compare the pH of the patients.
arterial blood gas parameters | During 28 days in the intensive care unit
  It was aimed to compare the base excess of the patients.
arterial blood gas parameters | During 28 days in the intensive care unit
  It was aimed to compare the lactate of the patients.
arterial blood gas parameters | During 28 days in the intensive care unit
  It was aimed to compare the partial oxygen pressure of the patients.

CONTACTS AND LOCATIONS:
Locations (1):
- Basaksehir Cam Sakura City Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] DesPrez K, McNeil JB, Wang C, Bastarache JA, Shaver CM, Ware LB. Oxygenation Saturation Index Predicts Clinical Outcomes in ARDS. Chest. 2017 Dec;152(6):1151-1158. doi: 10.1016/j.chest.2017.08.002. Epub 2017 Aug 16. PMID 28823812
- [Background] Chen WL, Lin WT, Kung SC, Lai CC, Chao CM. The Value of Oxygenation Saturation Index in Predicting the Outcomes of Patients with Acute Respiratory Distress Syndrome. J Clin Med. 2018 Aug 8;7(8):205. doi: 10.3390/jcm7080205. PMID 30096809
- [Background] Amato MB, Meade MO, Slutsky AS, Brochard L, Costa EL, Schoenfeld DA, Stewart TE, Briel M, Talmor D, Mercat A, Richard JC, Carvalho CR, Brower RG. Driving pressure and survival in the acute respiratory distress syndrome. N Engl J Med. 2015 Feb 19;372(8):747-55. doi: 10.1056/NEJMsa1410639. PMID 25693014
- [Result] ARDS Definition Task Force; Ranieri VM, Rubenfeld GD, Thompson BT, Ferguson ND, Caldwell E, Fan E, Camporota L, Slutsky AS. Acute respiratory distress syndrome: the Berlin Definition. JAMA. 2012 Jun 20;307(23):2526-33. doi: 10.1001/jama.2012.5669. PMID 22797452
- [Result] Bellani G, Laffey JG, Pham T, Fan E, Brochard L, Esteban A, Gattinoni L, van Haren F, Larsson A, McAuley DF, Ranieri M, Rubenfeld G, Thompson BT, Wrigge H, Slutsky AS, Pesenti A; LUNG SAFE Investigators; ESICM Trials Group. Epidemiology, Patterns of Care, and Mortality for Patients With Acute Respiratory Distress Syndrome in Intensive Care Units in 50 Countries. JAMA. 2016 Feb 23;315(8):788-800. doi: 10.1001/jama.2016.0291. PMID 26903337
- [Result] Sayed M, Riano D, Villar J. Novel criteria to classify ARDS severity using a machine learning approach. Crit Care. 2021 Apr 20;25(1):150. doi: 10.1186/s13054-021-03566-w. PMID 33879214
- [Result] Serpa Neto A, Deliberato RO, Johnson AEW, Bos LD, Amorim P, Pereira SM, Cazati DC, Cordioli RL, Correa TD, Pollard TJ, Schettino GPP, Timenetsky KT, Celi LA, Pelosi P, Gama de Abreu M, Schultz MJ; PROVE Network Investigators. Mechanical power of ventilation is associated with mortality in critically ill patients: an analysis of patients in two observational cohorts. Intensive Care Med. 2018 Nov;44(11):1914-1922. doi: 10.1007/s00134-018-5375-6. Epub 2018 Oct 5. PMID 30291378
- [Result] Asar S, Rahim F, Rahimi P, Acicbe O, Tontu F, Cukurova Z. Novel Oxygenation and Saturation Indices for Mortality Prediction in COVID-19 ARDS Patients: The Impact of Driving Pressure and Mechanical Power. J Intensive Care Med. 2024 Jun;39(6):595-608. doi: 10.1177/08850666231223498. Epub 2024 Jan 5. PMID 38179691
- [Result] Gattinoni L, Tonetti T, Cressoni M, Cadringher P, Herrmann P, Moerer O, Protti A, Gotti M, Chiurazzi C, Carlesso E, Chiumello D, Quintel M. Ventilator-related causes of lung injury: the mechanical power. Intensive Care Med. 2016 Oct;42(10):1567-1575. doi: 10.1007/s00134-016-4505-2. Epub 2016 Sep 12. PMID 27620287
- [Result] Asar S, Acicbe O, Cukurova Z, Hergunsel GO, Canan E, Cakar N. Bedside dynamic calculation of mechanical power: A validation study. J Crit Care. 2020 Apr;56:167-170. doi: 10.1016/j.jcrc.2019.12.027. Epub 2020 Jan 2. PMID 31931417